CLINICAL TRIAL: NCT00947076
Title: A Comparative Bioavailability Study of Fluoxetine Hydrochloride Capsules, 40 mg
Brief Title: To Demonstrate the Relative Bioavailability of Fluoxetine Hydrochloride Capsules, 40 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 005-49-11634
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Depression
Keywords: Antidepressant
MeSH Terms: conditions — Depression | interventions — Fluoxetine

ARMS (2):
- 1 (Experimental): Fluoxetine Hydrochloride Capsules, 40 mg (Geneva Pharmaceutical, Inc)
  Interventions: Drug: Fluoxetine Hydrochloride Capsules, 40 mg (Geneva Pharmaceutical, Inc)
- 2 (Active Comparator): Fluoxetine Hydrochloride Capsules, 40 mg (Prozac) (Eli Lilly)
  Interventions: Drug: Fluoxetine Hydrochloride Capsules, 40 mg (Prozac) (Eli Lilly)

INTERVENTIONS:
Drug: Fluoxetine Hydrochloride Capsules, 40 mg (Geneva Pharmaceutical, Inc)
  Arms: 1
Drug: Fluoxetine Hydrochloride Capsules, 40 mg (Prozac) (Eli Lilly)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of fluoxetine hydrochloride capsules, 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-02; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.